CLINICAL TRIAL: NCT00981214
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Pancreatic Enzyme Product (PEP) Microtabs in Pediatric Patients With Cystic Fibrosis and Exocrine Pancreatic Insufficiency
Brief Title: Study of Pancreatic Enzyme Product in Pediatric Participants With Cystic Fibrosis and Exocrine Pancreatic Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUR-1009-M
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: Cystic fibrosis; Exocrine Pancreatic Insufficiency; Zenpep-1009
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUR-1008 (APT-1008) (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008)

INTERVENTIONS:
Drug: EUR-1008 (APT-1008) — EUR-1008 (APT-1008) Microtabs contained in a capsule will be administered orally from Day 5 to Day 11 at an enzyme dose based on investigator's discretion, in dose stabilization period or the content of the capsule will be allowed to sprinkle on food, where necessary, followed by stabilized dose from Day 12 to Day 18 in treatment period, up to a maximum total dose of 10,000 lipase units per kilogram body weight per day (unit/kg/day).
  Other Names: ZENPEP®; Pancrelipase

SUMMARY:
This is an open-label study to evaluate the efficacy and safety of Aptalis' (formerly Eurand) pancreatic enzyme product (PEP) microtabs in pediatric participants under age 7 with cystic fibrosis (CF) and exocrine pancreatic insufficiency (EPI).

DETAILED DESCRIPTION:
The study sample will consist of evaluable participants, all of whom will be children younger than 7 years of age. Participants will receive EUR-1008 (APT-1008) Microtabs formulation. The study design involves a 4-day screening period, a 7-day dose stabilization period, and a 7-day treatment period (excluding an end-of-study evaluation).

The optimal dose of EUR-1008 (APT-1008) Microtabs, determined during the dose stabilization period, will be used during the treatment period. Participants are instructed to consume a predefined diet.

ELIGIBILITY:
Inclusion Criteria:

* Participants less than 7 years of age
* Participants who have pancreatic insufficiency documented by a fecal elastase level less than 100 micrograms per gram (mcg/g), or if not documented, the fecal elastase test must be done at the screening visit
* Participants who have a need of de novo treatment with pancreatic enzymes or be able to be switched from an existing treatment
* Participants who have a body mass index greater than the twenty fifth percentile for children 2 years and older
* Participants with a weight for height index greater than the twenty fifth percentile for children less than 2 years of age
* Participants with diagnosis of CF based upon the following criteria:

  * Have 2 clinical features consistent with CF and
  * Have either a genotype with 2 identifiable mutations consistent with CF or a sweat chloride concentration that is more than 60 milliequivalent per liter (mEq/L) by quantitative pilocarpine iontophoresis
* Participants who are clinically stable with no evidence of acute upper or lower respiratory tract infection

Exclusion Criteria:

* Participants with fibrosing colonopathy
* Participants allergic to pork or other porcine PEPs
* Participants with any respiratory condition that in the investigator's opinion would result in an intervention requiring hospitalization or intensive pulmonary treatment during the trial
* Participants with any acute systemic administration of an antibiotic for any reason in the previous 4 weeks; however, a low stable dose of an antibiotic (such as azithromycin 250 or 500 milligram [mg] up to 3 times per week) is allowed. Moreover, chronic treatment (that is, daily for at least 1 month) with an inhalatory antibiotic (for example, colistin, tobramycin, or ceftazidime) is allowed
* Participants who have hepatic insufficiency as defined by a history or presence of ascites, or a serum albumin level of less than 3.0 milligram per deciliter (mg/dL), or coagulopathy with an international normalized ratio that is greater than 1.7
* Participants with hyperuricemia or hyperuricosuria
* Participants participating in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to screening visit
* Participants with history of or current screening evaluation of hyperglycemia as defined by an 8-hour fasting serum glucose equivalent to 126 mg/dL or more, or of cystic-fibrosis-related diabetes as determined according to the Cystic Fibrosis Foundation (CFF) Consensus Conference of January 1999 (Section IX Part II), that is:

  * Fasting Blood Glucose (FBG) greater than126 mg/dl (7.0 milli mole [mM]) on two or more occasions
  * FBG greater than 126 mg/dl (7 .0 mM) plus casual (without regard to time of day or last meal consumed) glucose level greater than200 mg/dl (11.1 mM)
  * Casual (previously called random) glucose levels greater than 200 mg/dl (11.1 mM) on two or more occasions with symptoms
* Participants with any solid organ transplant or surgery affecting the bowel
* Participants using an enzyme preparation in excess of 10,000 lipase units/kg/day
* Participants with an acute dose of any steroid in the previous 2 weeks; however, low chronic doses of a steroid (less 0.5 mg/kg every other day) will be allowed
* Participants with any condition that would, in the investigator's opinion, limit the patient's ability to complete the study
* Participants with history of or current screening determination of distal ileal obstruction syndrome (DIOS), or any clinical signs and symptoms suggestive of DIOS (that is, constipation, abdominal pain, anorexia, early satiety, recurrent vomiting and palpable fecal mass) on physical examination
* Participants who are unable to discontinue excluded concomitant medications over the course of the study

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2006-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (14):
- United States (14):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital - Oakland, Oakland, California
  - Stanford University Medical Center, Palo Alto, California
  - Children's Hospital of San Diego, San Diego, California
  - University of Florida College of Medicine, Gainsville, Florida
  - Nemours Childrens Clinic, Jacksonville, Florida
  - Childrens Memorial Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Cystic Fibrosis Center, Ann Arbor, Michigan
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - West Virginia Health Sciences Center, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) Microtabs contained in a capsule was administered orally from Day 5 to Day 11 at an enzyme dose based on investigator's discretion, in dose stabilization period or the content of the capsule was allowed to sprinkle on food, where necessary, followed by stabilized dose from Day 12 to Day 18 in treatment period, up to a maximum total dose of 10,000 lipase units per kilogram body weight per day (unit/kg/day).
Period: Overall Study
Arm/Group | EUR-1008 (APT-1008)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.9 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Percentage of Participants Who Were Responders [Number; unit: percentage of participants] — Responders were defined as those participants without steatorrhea (defined as less than 30 percent (%) fecal fat content) and without signs and symptoms of malabsorption at baseline (under currently available pancreatic enzyme products taken during the screening period).
  percentage of participants | 52.6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Responders After 1 Week of Treatment With Study Medication
Description: Responders were defined as those participants without steatorrhea (defined as less than 30 percent (%) fecal fat content) and without signs and symptoms of malabsorption after 1 week of treatment with study medication.
Time Frame: Day 11
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
percentage of participants | 68.4 [43.4 to 87.4]

2. Secondary Outcome: Change From Baseline in Weight at Day 12, 19
Time Frame: Baseline, Day 12, 19
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
kilogram
  Baseline | 16.60 (3.843)
  Change at Day 12 | 0.15 (0.401)
  Change at Day 19 | 0.03 (0.529)

3. Secondary Outcome: Mean Daily Number of Stools
Description: Mean daily number of stools of each participant was calculated from frequency of stools by the participant per day. Mean daily number of stools at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period), Day 12 up to Day 18 (treatment period)
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Error); unit: stools per day
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
stools per day
  Baseline | 1.82 (0.787)
  Dose stabilization period | 1.64 (0.722)
  Treatment period | 1.45 (0.548)

4. Primary Outcome: Percentage of Participants Who Were Responders After 2 Weeks of Treatment With Study Medication
Description: Responders were defined as those participants without steatorrhea (defined as less than 30% fecal fat content) and without signs and symptoms of malabsorption after 2 weeks of treatment with study medication.
Time Frame: Day 18 (end of treatment)
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
percentage of participants | 57.9 [33.5 to 79.7]

5. Secondary Outcome: Percentage of Stool Categorized by Consistency
Description: Stool consistency was categorized as hard, formed/normal, soft, watery or overt diarrhea. Percentage of stools of a specific consistency of each participant was calculated as the number of stools with a specific consistency relative to the total number of stools during the collection period. Mean percentage of stool with specific consistency at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period) and Day 12 up to Day 18 (treatment period)
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
percentage of stools
  Hard: Baseline | 5.45 (15.782)
  Hard: Dose stabilization period | 4.59 (12.694)
  Hard: Treatment period | 3.78 (8.624)
  Formed/Normal: Baseline | 59.46 (37.956)
  Formed/Normal: Dose stabilization period | 58.20 (33.675)
  Formed/Normal: Treatment period | 59.38 (35.671)
  Soft: Baseline | 30.18 (33.382)
  Soft: Dose stabilization period | 32.32 (28.283)
  Soft: Treatment period | 33.15 (31.460)
  Watery: Baseline | 4.54 (8.339)
  Watery: Dose stabilization period | 3.03 (6.988)
  Watery: Treatment period | 3.16 (6.561)
  Overt Diarrhea: Baseline | 0.38 (1.639)
  Overt Diarrhea: Dose stabilization period | 1.86 (8.097)
  Overt Diarrhea: Treatment period | 0.53 (2.294)

6. Secondary Outcome: Mean Number of Abdominal Symptoms: Bloating
Description: Bloating is swelling of the intestinal tract caused by excessive gas formation. Symptoms of bloating were classified by severity as mild (no impairment of daily activities), moderate (slight impairment of daily activities), or severe (unable to perform daily activities). Mean number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Mean number of symptoms at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period), Day 12 up to Day 18 (treatment period)
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: bloatings per day
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
bloatings per day
  Mild: Baseline | 0.11 (0.326)
  Mild: Dose stabilization period | 0.14 (0.391)
  Mild: Treatment period | 0.08 (0.230)
  Moderate: Baseline | 0.06 (0.159)
  Moderate: Dose stabilization period | 0.02 (0.098)
  Moderate: Treatment period | 0.01 (0.029)
  Severe: Baseline | 0.04 (0.172)
  Severe: Dose stabilization period | 0.00 (0.000)
  Severe: Treatment period | 0.00 (0.000)

7. Secondary Outcome: Mean Number of Abdominal Symptoms: Flatulence
Description: Flatulence is presence of excessive gas in the digestive tract. Symptoms of flatulence was classified by severity as mild (no impairment of daily activities), moderate (slight impairment of daily activities), or severe (unable to perform daily activities). Mean number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Mean number of symptoms at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period), Day 12 up to Day 18 (treatment period)
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: flatulences per day
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
flatulences per day
  Mild: Baseline | 0.13 (0.262)
  Mild: Dose stabilization period | 0.20 (0.283)
  Mild: Treatment period | 0.08 (0.215)
  Moderate: Baseline | 0.06 (0.109)
  Moderate: Dose stabilization period | 0.06 (0.204)
  Moderate: Treatment period | 0.00 (0.000)
  Severe: Baseline | 0.04 (0.119)
  Severe: Dose stabilization period | 0.02 (0.045)
  Severe: Treatment period | 0.09 (0.393)

8. Secondary Outcome: Mean Number of Pain Symptoms
Description: Symptoms of pain was classified by severity as mild (no impairment of daily activities), moderate (slight impairment of daily activities), or severe (unable to perform daily activities). Mean number of symptoms of specific severity for each participant was calculated from frequency of symptoms by the participant per day. Mean number of symptoms at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period), Day 12 up to Day 18 (treatment period)
Population: Analysis population set included all participants who received at least 1 dose of study.
Measure: Mean (Standard Deviation); unit: pain symptoms per day
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
pain symptoms per day
  Mild: Baseline | 0.09 (0.210)
  Mild: Dose stabilization period | 0.14 (0.321)
  Mild: Treatment period | 0.07 (0.204)
  Moderate: Baseline | 0.04 (0.118)
  Moderate: Dose stabilization period | 0.08 (0.204)
  Moderate: Treatment period | 0.00 (0.000)
  Severe: Baseline | 0.00 (0.000)
  Severe: Dose stabilization period | 0.05 (0.201)
  Severe: Treatment period | 0.00 (0.000)

9. Secondary Outcome: Physician's and Parent's or Legal Guardians Assessment of Improvement in Clinical Symptoms
Description: Clinical symptoms of exocrine pancreatic insufficiency (EPI) were assessed by the physician and parent or guardian to determine if the participant showed improvement in symptoms of EPI at end of study after the dose stabilization period. EPI is a syndrome characterized by clinical symptoms of poor absorption of fats, proteins, and to a lesser extent, carbohydrates, which manifests primarily in patients with cystic fibrosis. Number of participants with improvement in clinical symptoms was reported.
Time Frame: Day 19 (end of study)
Population: Analysis population set included all participants who received at least 1 dose of study.
Measure: Number; unit: participants
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
participants
  Physician assessment | 7
  Parent/guardian assessment | 9

10. Secondary Outcome: Percentage of Blood in Stool
Description: Mean percentage of stools with blood at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period), Day 12 up to Day 18 (treatment period)
Population: Analysis population set included all participants who received at least 1 dose of study.
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
percentage of stools
  Baseline | 0 (0)
  Dose stabilization period | 0 (0)
  Treatment period | 0 (0)

11. Secondary Outcome: Percentage of Stool With Visible Oil or Grease
Description: Mean percentage of oil or grease at each period for total participants was summarized.
Time Frame: Baseline, Day 5 up to Day 11 (dose stabilization period), Day 12 up to Day 18 (treatment period)
Population: Analysis population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 19
percentage of stools
  Baseline | 11.10 (14.433)
  Dose stabilization period | 8.98 (11.879)
  Treatment period | 4.73 (7.722)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 19
Description: Adverse event (AE) was defined as any untoward medical occurrence regardless of causal relationship to study medication. Serious AE was any event that resulted in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity, or was a congenital anomaly/birth defect.
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) Microtabs contained in capsule was administered orally or sprinkled on food. When required, from Day 5 to Day 11 at an enzyme dose based on investigator's discretion, in dose stabilization period or allowed to sprinkle on food, where necessary, followed by stabilized dose from Day 12 to Day 18 in treatment period, up to a maximum total dose of 10,000 lipase units per kilogram body weight per day (unit/kg/day).
Arm/Group | EUR-1008 (APT-1008)
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 13/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EUR-1008 (APT-1008) (N=19)
Upper respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EUR-1008 (APT-1008) (N=19)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lacrimation increased (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Steatorrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3

LIMITATIONS AND CAVEATS:
Protocol amendment 4 extended screening period to 14 days, but this period not included in result as all participants started treatment prior to site Institutional Review Board approval of protocol amendment 4, this did not affect study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.